CLINICAL TRIAL: NCT04972058
Title: Philippine Neurological Association One Database - Stroke
Acronym: PNA1DB-Stroke
Status: Completed | Type: Observational
Sponsor: Philippine Neurological Association (Other)
Responsible Party: Sponsor
Other Study IDs: PNA1DB-Stroke
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Transient Ischemic Attack; Ischemic Stroke; Intracerebral Hemorrhage; Subarachnoid Hemorrhage; Cerebral Venous Thrombosis
MeSH Terms: conditions — Ischemic Attack, Transient; Ischemic Stroke; Cerebral Hemorrhage; Subarachnoid Hemorrhage; Intracranial Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a pragmatic, multi-center, prospective, observational, non-interventional study and standing database of patients hospitalized for transient ischemic attack (TIA) or stroke in the 11 accredited adult neurology training institutions in the Philippines. Data will be collected from each patient while admitted in the hospital and until hospital discharge. Data collection for this study will span 3 years from study initiation, after which the utility of an extension or a re-implementation of the study will be assessed.

DETAILED DESCRIPTION:
Primary objective is to prospectively collect data on demographics, medical history, in-hospital management, and outcomes among patients with first or recurrent TIA or ischemic or hemorrhagic stroke admitted in accredited adult neurology training institutions in the Philippines.

Secondary objectives are:

1. To determine the in-patient case load of first and recurrent TIA and stroke.
2. To determine the profile of patients admitted for first or recurrent TIA or stroke.
3. To determine the types of diagnostic and therapeutic management received by patients with first or recurrent TIA or stroke.
4. To determine the outcomes of patients with first or recurrent TIA or stroke at the time of hospital discharge.
5. To evaluate factors that predict outcome among patients with first or recurrent TIA or stroke.
6. To assess and audit the overall quality of care received by patients admitted for first or recurrent TIA or stroke.
7. To perform other future analyses, sanctioned by the Philippine Neurological Association (PNA), that may improve knowledge on the care of patients with first and/or recurrent TIA or stroke.

All eligible patients will be assigned a study identification (ID) number and included in the site log kept confidentially in each site. Corresponding anonymized data on demographics, medical history, stroke sub-type, in-hospital management and discharge outcomes will be collected from each patient and entered in the database using a secure online data collection tool.

Collective data will be extracted, summarized, and analyzed for the secondary objectives every year with oversight provided by the Philippine Neurological Association.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of first or recurrent TIA, ischemic or hemorrhagic stroke, or cerebral venous thrombosis (CVT)
2. 18 years old or older
3. Admitted in the participating hospital
4. If required by the institutional review board/ethics committee, signed or verbal informed consent for participation in the study from the patient or a legal representative

Exclusion Criteria:

1. Patients with previous TIA or stroke who are admitted to the hospital for medical conditions other than an acute stroke, e.g., patient with non-acute stroke admitted for pneumonia, rehabilitation, or procedures, such as gastric tube insertion, etc.
2. Any condition which, in the study investigator's opinion, may jeopardize the patient by his/her participation in this study or affect the validity of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted at the participating sites fulfilling all inclusion and none of the exclusion criteria are eligible to be included.
Sampling Method: Non-Probability Sample
Enrollment: 14800 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
In-hospital caseload | 3 years
  Number of TIA and stroke cases admitted in participating sites.

SECONDARY OUTCOMES:
In-hospital diagnostic procedure (brain scan) | From admission to discharge, may be up to 1 month
  Rate of performance of brain scan.
In-hospital diagnostic procedures (electrocardiogram) | From admission to discharge, may be up to 1 month
  Rate of performance of electrocardiogram.
In-hospital diagnostic procedures (echocardiogram) | From admission to discharge, may be up to 1 month
  Rate of performance of echocardiogram.
In-hospital diagnostic procedures (cerebral vascular studies) | From admission to discharge, may be up to 1 month
  Rate of performance of any cerebral vascular study.
In-hospital therapeutic management (thrombolysis) | From admission to discharge, may be up to 1 month
  Rate of treatment with thrombolysis (intravenous and/or endovascular).
In-hospital therapeutic management (anti-thrombotics) | From admission to discharge, may be up to 1 month
  Rate of treatment with any anti-thrombotic (anti-platelet and/or anti-coagulant).
In-hospital therapeutic management (rehabilitation) | From admission to discharge, may be up to 1 month
  Rate of rehabilitation (physical therapy and/or occupational therapy and or speech therapy).
In-hospital complications from TIA or stroke | From admission to discharge, may be up to 1 month
  Rate of complications arising from TIA or stroke.
Vital status at hospital discharge | At discharge, may be up to 1 month
  Alive or dead
Functional status at hospital discharge | At discharge, may be up to 1 month
  modified Rankin Scale
Neurological status at hospital discharge | At discharge, may be up to 1 month
  National Institute of Health Stroke Scale

CONTACTS AND LOCATIONS:
Overall Officials: Robert N Gan, MD, Study Chair — Philippine Neurological Association
Locations (11):
- Philippines (11):
  - Baguio General Hospital and Medical Center, Baguio City, Benguet
  - Chong Hua Hospital, Cebu City
  - Makati Medical Center, Makati City
  - Jose R. Reyes Memorial Medical Center, Manila
  - University of Santo Tomas Hospital, Manila
  - University of the Philippines - Philippine General Hospital, Manila
  - The Medical City, Pasig
  - East Avenue Medical Center, Quezon City
  - Quirino Memorial Medical Center, Quezon City
  - St. Luke's Medical Center (QC, BGC), Quezon City
  - University of the East - Ramon Magsaysay Memorial Medical Center, Quezon City

REFERENCES:
- [Derived] Philippine Neurological Association One Database - Stroke, Disease Study Management Group. Multicentre collection of uniform data on patients hospitalised for transient ischaemic attack or stroke in the Philippines: the Philippine Neurological Association One Database-Stroke (PNA1DB-Stroke) protocol. BMJ Open. 2022 May 24;12(5):e055954. doi: 10.1136/bmjopen-2021-055954. PMID 35613760